CLINICAL TRIAL: NCT04245748
Title: Determining Optimal Treatment Sequences in Anxious Depression (DOTS-AD)
Acronym: DOTS-AD
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Cincinnati (Other)
Responsible Party: Principal Investigator, Jeffrey Strawn, MD, Associate Professor of Psychiatry & Pediatrics, Director, Anxiety Disorders Research Program, University of Cincinnati
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Strawn DOTS-AD
Record Dates: First submitted 2020-01-27; First posted 2020-01-29 (Actual); Last update posted 2024-08-29 (Actual); Status verified 2024-08

CONDITIONS: Anxious Depression; Depression
Keywords: Anxious Depression
MeSH Terms: conditions — Depression | interventions — Escitalopram; Duloxetine Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Escitalopram (Active Comparator): Adaptively randomized, double-blind treatment with escitalopram for 11 weeks in Phase 1. Non-remitting patients will be randomized in Phase 2 to adjunctive clonazepam or pregabalin for 8 weeks. Additionally, adults who are already treated with escitalopram or citalopram for at least 6 weeks prior to screening, may enter Phase 2 and be randomized to adjunctive clonazepam or pregabalin for 8 weeks.
  Interventions: Drug: Escitalopram
- Duloxetine (Active Comparator): Adaptively randomized, double-blind treatment with duloxetine for 11 weeks in Phase 1. Non-remitting patients will be randomized in Phase 2 to adjunctive clonazepam or pregabalin for 8 weeks. Additionally, adults who are already treated with duloxetine for at least 6 weeks prior to screening, may enter Phase 2 and be randomized to adjunctive clonazepam or pregabalin for 8 weeks.
  Interventions: Drug: Duloxetine

INTERVENTIONS:
Drug: Escitalopram — Escitalopram, a SSRI, commercially known as LexaproTM, is commonly prescribed for anxiety disorders and is FDA-approved for acute and maintenance treatment of MDD and GAD.
  Other Names: Lexapro
  Arms: Escitalopram
Drug: Duloxetine — Duloxetine, a SNRI, commercially known as CymbaltaTM, is FDA-approved for the treatment of GAD, MDD, diabetic peripheral neuropathic pain, fibromyalgia, and chronic musculoskeletal pain in adults.
  Other Names: Cymbalta
  Arms: Duloxetine

SUMMARY:
Acute, double-blind, adaptively randomized treatment with duloxetine or escitalopram, followed by double-blind, randomized adjunctive treatment with clonazepam or pregabalin for persistent symptoms.

DETAILED DESCRIPTION:
The study will consist of 2 phases (Figure 1). Eighty-four adults will be enrolled in Phase 1 and will be adaptively randomized (initially 1:1) to acute, double-blind treatment with escitalopram or duloxetine for 11 weeks. Remission status will be determined at week 10. Remitting patients (CGI-S ≤2) will resume treatment as usual, which may consist of outpatient referral. Non-remitting patients (CGI-S ≥3), will continue into Phase 2 and will be randomized to adjunctive clonazepam or pregabalin for 8 weeks. Twenty adults treated with escitalopram (or its racemic equivalent, citalopram) or duloxetine for ≥6 weeks (at screening) will be enrolled into Phase 2 and will be randomized to receive adjunctive clonazepam or pregabalin for 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Written, informed consent.
* Patients must be fluent in the English.
* 18 to 50 years of age, inclusive, at Visit 1.
* Patients must meet DSM-5 criteria for generalized, social and/or separation anxiety disorder and/or panic disorder, confirmed by the MINI.99 Patients may also meet criteria for persistent depressive disorder or major depressive disorder however, these may not be the primary focus of treatment.
* HAM-A score ≥20 at Visits 1 and 2.
* Clinical Global Impressions- Severity (CGI-S) score ≥4 at Visits 1 and 2.
* No clinically significant abnormalities on physical examination and EKG.
* Negative pregnancy test at Visit 1 in females.
* Negative urine drug screen at Visit 1.
* Sexually active patients must practice a reliable method of contraception (Section 15.0) that will continue for the duration of the study and for a minimum of 30 days following the end of study participation. Reliable methods of contraception are defined below; other forms of contraceptives (pharmacological and/or non-pharmacological) are not accepted:

  1. Surgical sterilization
  2. Oral contraceptives (e.g. estrogren-progestin combination or progestin)
  3. Transdermally-delivered contraceptives (e.g., Ortho-Evra), depot injections (e.g., Depo-Provera)
  4. Vaginal contraceptive ring (e.g., NuvaRing), contraceptive implants (e.g., Implanon, Norplant II/Jadelle)
  5. An intrauterine device
  6. Diaphragm plus condom.
* For patients directly enrolling into Phase 2: treatment with escitalopram (or its racemic equivalent citalopram) or duloxetine for ≥6 weeks, at time of screening.

Exclusion Criteria:

* DSM-5 diagnosis other than generalized anxiety, social anxiety, separation anxiety or panic disorder(s) that is the primary focus of treatment.
* A history of intellectual disability.
* Suicide risk as determined by either: (1) any suicide attempt within the past 6 months and/or (2) significant risk at Visit 1 (Screening) or Visit 2 (Baseline), as judged by the Investigator.
* Allergy, intolerance, non-response or hypersensitivity to escitalopram, duloxetine, pregabalin or clonazepam.
* Subjects taking other medications that require a taper or washout of more than 5 days.
* Patients who have initiated/terminated psychotherapy/behavior therapy within 1 month before Visit 2 (Baseline) will be excluded; if the patient is engaged in psychotherapy, it must have been stable for 1 month prior to baseline.
* A clinically-significant medical illness.
* QTc >450 in males or >460 in females (prolonged QTc based on American Heart Association recommendations for Standardization and Interpretation of the EKG100
* Alcohol or substance use disorder within 6 months of baseline (nicotine use is permitted).
* Positive urine pregnancy test/pregnancy or breast feeding.
* A positive urine drug screen.
* Patients who are unable to swallow capsules.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 84 (Estimated)
Dates: Start 2020-03-01 (Actual); Primary Completion 2025-07-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Hamilton Anxiety Rating Scale (HAM-A) total score | Week 2 to 20
  The HAM-A rating scale is a test of 14 items measuring the severity of anxiety symptoms. Each item is rated on a 5-point ordinal scale, ranging from 0 (not present) to 4 (severe). Total scores range from 0 to 56. A lower score is favorable.
Change from Baseline in the Clinical Global Impression of Severity (CGI-S) | Week 2 to 20
  CGI-S is a seven point scale where 1=Normal and 7=Among the most extremely ill patients.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey R Strawn, MD, FAACAP, Principal Investigator — University of Cincinnati
Locations (1):
- University of Cincinnati, Department of Psychiatry & Behavioral Neuroscience, Cincinnati, Ohio, United States